CLINICAL TRIAL: NCT03362710
Title: Evaluation du Risque Vasculaire Par Mesures Non Invasives en Soins Primaires.
Brief Title: Simplified and Easy Detection of Arterial Disease in Nursing Homes
Acronym: First-SEDAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A02635-48
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2020-08

CONDITIONS: Artery Disease, Peripheral
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PAD patients (Experimental): Patients referred for an arterial doppler assessment of lower limbs will be included.
  Intervention is a series of examination, followed by the measurement of the ABI and an arterial echo-doppler of the lower limbs +/- transcutaneous oxygen pressure measurements in case of suspected critical limb ischemia.
  A technician will perform the evaluation with simplified tools blinded to the results of vascular specialised investigations
  Interventions: Diagnostic Test: simplified tools

INTERVENTIONS:
Diagnostic Test: simplified tools — 1. Skin temperature on the back of the foot with infra-red thermometry
  2. Toe saturometry
  3. ABI with an automatic sphygmomanometry
  4. Skin Recoloration time at the foot

SUMMARY:
Peripheral artery disease (PAD) affects mainly elderly patients. The ankle brachial index (ABI) and ultrasound imaging are the standard diagnostic tools in PAD diagnostic and severity estimation. Measurements are generally performed by a vascular physician. However, access to medical specialist is becoming increasingly difficult with long waiting times while the aging of the population increases, while most of these patients are seen by the general practitioner.

To date, there is a lot of data in the literature on the value of using various ambulatory devices in the diagnosis and severity estimation of PAD but studied one by one.

The investigators propose to compare the measurements made by a series of simple non-invasive ambulatory tools with the measurements performed by the vascular specialist. The investigators wish to demonstrate that a series of simple and economical tools, available to paramedical health professionals can diagnose PAD and evaluate ts severity the reducing the direct and indirect associated costs.

DETAILED DESCRIPTION:
Patients referred for an arterial vascular investigations of the lower limbs will be included.

After signing the consent, all included patients will be assessed by the examination series, among which ABI measurement and an arterial Doppler ultrasound of the lower limbs +/- transcutaneous oxygen pressure recording in case of suspected critical limb ischemia. Following the visit patients will be classified as have or not PAD and in case of PAD classified for the severity of PAD on the basis of the investigation results.

Blinded to the results of the vascular laboratory test, a technician will:

Measure ABI with an automatic sphygmomanometer.

Examination series:

1. Skin temperature on the back of the foot with infra-red thermometry
2. Toe saturometry
3. ABI with an automatic sphygmomanometry
4. Skin Recoloration time at the foot

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for arterial assessment of the lower limbs as part of a screening or follow-up of PAD
* Patients without contraindications for all non-invasive measures
* Age superior to 18 years
* Affiliated patients of a social security scheme
* Patients who have signed informed consent.

Exclusion Criteria:

* Patients protected by law
* Patients unable to understand the objectives or instructions of the study
* Patients in an exclusion period relative to another biomedical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Performance of non-invasive measurements | 1 hour
  Performance of the score will be studied with the receiver operating characteristic (ROC) approach and multivariate analysis using echo-doppler and transcutaneous oxymetry results as references for PAD severity classification standard

CONTACTS AND LOCATIONS:
Overall Officials: Samir HENNI, MD,PhD, Principal Investigator — UH Angers
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No